CLINICAL TRIAL: NCT02696278
Title: Hummus for Health: Dietary Quality and Health Outcomes in Toddlers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study product voluntarily recalled by sponsor. Listeria identified at the manufacturing facility (not in tested finished product).
Sponsor: Baylor College of Medicine (Other)
Collaborators: Sabra Dipping Company, LLC (Other)
Responsible Party: Principal Investigator, Sheryl Hughes, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 47364-I; H-38273 (Other: Baylor College of Medicine)
Record Dates: First submitted 2015-12-31; First posted 2016-03-02 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Obesity
Keywords: gut microbiota; obesity; toddlers; fiber; unsaturated fats
MeSH Terms: conditions — Obesity | interventions — Vegetables

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hummus and vegetables (Experimental): Children will receive a lesson about vegetables and hummus and vegetables as part of their daily snack.
  Interventions: Other: Lesson about vegetables; Other: Vegetables; Other: Hummus
- Vegetables only (Experimental): Children will receive a lesson about vegetables and vegetables as part of their daily snack.
  Interventions: Other: Lesson about vegetables; Other: Vegetables

INTERVENTIONS:
Other: Lesson about vegetables — During the introductory period, children will receive a lesson about vegetables 3 days a week for 3 weeks.
Other: Vegetables — During the introductory period, children will be served vegetables 3 days a week for 3 weeks during snack time at their daycare center. During the intervention period, children will receive vegetables everyday for 3 weeks during snack time at their daycare center.
Other: Hummus — During the introductory period, children will be served hummus, depending on their group assignment, 3 days a week for 3 weeks during snack time at their daycare center. During the intervention period, children will receive hummus, depending on their group assignment, everyday for 3 weeks during snack time at their daycare center.
  Arms: Hummus and vegetables

SUMMARY:
The goal of this study is to examine the effect of increasing children's intake of fiber and unsaturated fat, through daily servings of hummus and vegetables, on their microbiome profile.

DETAILED DESCRIPTION:
Population: The investigators will recruit 104 children ages 12-24 months from daycare centers in the Houston and surrounding areas.

Study design: The study will be conducted at daycare centers and will consist of three phases - a 'lead in period' (two weeks) where baseline measurements will be taken followed by an 'Introductory period' (three weeks) where the new food will be introduced on three days during snack time for three weeks. The introductory phase will be followed by the 'intervention period' (three weeks) where children will receive daily servings of hummus and vegetables.

Lead in period (two weeks): Two 24-hour dietary recalls will be conducted on each child (parent-report); one 24-hour dietary recall (over a weekend) will be conducted on each parent (self-report). Three dirty diapers will be collected within the time span of a week for microbiome analysis.

Introductory period (three weeks): Since children typically take several introductions of a new food to accept it, and the investigators wish to ensure a high acceptance of hummus, the investigators will spend three weeks introducing the food. The food will be provided on three days during snack time for three weeks. Prior to introducing the food, children will receive a 'lesson' involving information about vegetables using a combination of songs, rhymes and craft activities. Following the lesson, hummus and vegetables will be provided in the hummus group; vegetables only in the control group. Hummus will be provided in a pre-packaged 2 ounce serving cup; vegetables will conform to age-appropriate servings designated by the American Academy of Pediatrics (AAP) and will consist of soft vegetables (e.g., winter squash) and lightly steamed, but chilled, hard vegetables (e.g., carrots, broccoli).

Intervention period (three weeks): Similar to the introductory period, a serving of either hummus and vegetables or vegetables only will be provided to the children during snack time. The food will be provided daily for three weeks. In the final week of the intervention period, two 24-hour dietary recalls (one weekday and one weekend) will be conducted on the child (parent-report). In addition, one weekend 24-hour dietary recall will be conducted on the parent (self-report). Three dirty diapers will be collected on the child during the final week for microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 12 and 24 month old.
* Children attending daycare at least 3 days a week.
* Children with a parental-report of being hummus-naive.

Exclusion Criteria:

* Any child following a specific dietary regimen or that has religious restrictions or food allergies that may affect food consumption.
* Children with parent-reported antibiotic use in the previous 6 months.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 139 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Children's Healthy Eating Index total score | 8 weeks
  Parent-report of 24-hour dietary recalls of the child's consumption will be used for this measure.
Children's microbiome profile | 8 weeks
  For this measure stool samples from the children will be collected.
Children's daily consumption of greens and beans | 8 weeks
  Parent-report of 24-hour dietary recalls of the child's consumption will be used for this measure.
Children's daily consumption of vegetables | 8 weeks
  Parent-report of 24-hour dietary recalls of the child's consumption will be used for this measure.
Children's daily consumption of unsaturated fats | 8 weeks
  Parent-report of 24-hour dietary recalls of the child's consumption will be used for this measure.

SECONDARY OUTCOMES:
Parent's Healthy Eating Index total score | 8 weeks
  Self-report of 24-hour dietary recalls of the parent's consumption will be used for this measure.
Parent's daily consumption of greens and beans | 8 weeks
  Self-report of 24-hour dietary recalls of the parent's consumption will be used for this measure.
Parent's daily consumption of vegetables | 8 weeks
  Self-report of 24-hour dietary recalls of the parent's consumption will be used for this measure.
Parent's daily consumption of unsaturated fats | 8 weeks
  Self-report of 24-hour dietary recalls of the parent's consumption will be used for this measure.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O Hughes, PhD, Principal Investigator — Baylor College of Medicine; Alexis Frazier-Wood, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arlinghaus KR, Vollrath K, Hernandez DC, Momin SR, O'Connor TM, Power TG, Hughes SO. Authoritative parent feeding style is associated with better child dietary quality at dinner among low-income minority families. Am J Clin Nutr. 2018 Oct 1;108(4):730-736. doi: 10.1093/ajcn/nqy142. PMID 30169719